CLINICAL TRIAL: NCT02258659
Title: An Exploratory Pilot Study of Nab-paclitaxel Based Induction Chemotherapy Followed by Response-Stratified Locoregional Therapy for Patients With Stage III and IV HPV-Related Oropharyngeal Cancer - the OPTIMA HPV Trial
Brief Title: Nab-paclitaxel and Carboplatin Followed by Response-Based Local Therapy in Treating Patients With Stage III or IV HPV-Related Oropharyngeal Cancer
Acronym: OPTIMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-0639; NCI-2014-01867 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB14-0639 (Other: University of Chicago); P30CA014599 (NIH)
Record Dates: First submitted 2014-09-19; First posted 2014-10-07 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Human Papilloma Virus Infection; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Papillomavirus Infections; Squamous Cell Carcinoma of Head and Neck | interventions — Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Carboplatin; Radiotherapy; Radiation; Paclitaxel; Fluorouracil; Hydroxyurea; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (radiation therapy alone) (Experimental): Patients undergo radiation therapy once daily for weeks.
  Interventions: Drug: paclitaxel albumin-stabilized nanoparticle formulation; Drug: carboplatin; Radiation: radiation therapy; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment
- Group B (combination chemotherapy, low-dose radiation therapy) (Experimental): Patients receive hydroxyurea PO BID on days 0-5, fluorouracil IV continuously on days 1-5, and paclitaxel IV over 60 minutes on day 1. Patients also receive low-dose radiation therapy BID on days 1-5. Treatment repeats every 14 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: paclitaxel albumin-stabilized nanoparticle formulation; Drug: carboplatin; Radiation: radiation therapy; Drug: paclitaxel; Drug: fluorouracil; Drug: hydroxyurea; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment
- Group C (combination chemotherapy, high-dose radiation) (Experimental): Patients receive hydroxyurea PO BID on days 0-5, fluorouracil IV continuously on days 1-5, and paclitaxel IV over 60 minutes on day 1. Patients also receive standard-dose radiation therapy BID on days 1-5. Treatment repeats every 14 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.*
  *NOTE: At the discretion of the PI, patients may receive cisplatin IV over 1-3 hours every 3 weeks during radiation therapy instead of paclitaxel and undergo daily radiation therapy.
  Interventions: Drug: paclitaxel albumin-stabilized nanoparticle formulation; Drug: carboplatin; Radiation: radiation therapy; Drug: paclitaxel; Drug: fluorouracil; Drug: hydroxyurea; Drug: cisplatin; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IV
  Other Names: ABI-007; nab paclitaxel; nab-paclitaxel; nanoparticle albumin-bound paclitaxel
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
  Arms: Group B (combination chemotherapy, low-dose radiation therapy); Group C (combination chemotherapy, high-dose radiation)
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
  Arms: Group B (combination chemotherapy, low-dose radiation therapy); Group C (combination chemotherapy, high-dose radiation)
Drug: hydroxyurea — Given PO
  Other Names: HU; HYD; Hydrea; Hydroxycarbamide; Hydurea
  Arms: Group B (combination chemotherapy, low-dose radiation therapy); Group C (combination chemotherapy, high-dose radiation)
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
  Arms: Group C (combination chemotherapy, high-dose radiation)
Other: laboratory biomarker analysis — Correlative studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This phase II trial studies nab-paclitaxel (paclitaxel albumin-stabilized nanoparticle formulation) and carboplatin followed by response-based local therapy in treating patients with stage III or IV human papillomavirus (HPV)-related oropharyngeal cancer. Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, carboplatin, hydroxyurea, fluorouracil, paclitaxel, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them spreading. Radiation therapy uses high energy x rays to kill tumor cells. Giving nab-paclitaxel and carboplatin before chemoradiation may make the tumor smaller and reduce the amount of chemotherapy and radiation therapy needed. Assigning chemotherapy and radiation therapy based on response (response-based therapy) and giving patients who are responding well lower doses of treatment may help reduce the occurrence of side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 2-year progression-free survival (PFS).

SECONDARY OBJECTIVES:

I. Clinical complete response rate (nab-paclitaxel based induction, compared to European Prospective Investigation into Cancer and Nutrition [EPIC] induction [paclitaxel based]).

II. Response rate (nab-paclitaxel based induction, compared to EPIC induction [paclitaxel based]).

III. Proportion of patients with >= 50% shrinkage by Response Evaluation Criteria In Solid Tumors (RECIST) (nab-paclitaxel based induction, compared to EPIC induction, paclitaxel based).

IV. Toxicity (nab-paclitaxel based induction, compared to EPIC induction [paclitaxel based]).

V. To assess swallowing function and speech at 6 months (mos) and 12 mos post therapy.

VI. To determine the rates of late toxicity with chemoradiation following surgery as determined by xerostomia, dental decay, osteroradionecrosis, G-tube dependency, tracheostomy placement and dysphagia.

VII. 2-year overall survival (OS) in patients treated on the Low-Risk, Intermediate-Risk Arm, and High-Risk Arms.

VIII. 2-year PFS in patients treated on the Low-Risk, Intermediate-Risk Arm, and High-Risk Arms - early and late toxicities.

IX. Evaluate need for post radiotherapy/chemoradiotherapy (RT/CRT) surgery on low- and intermediate-risk arms based on response from induction chemotherapy.

X. Evaluate in a descriptive manner the role of transoral robotic surgery (TORS) resection/lymph node dissection (LND) when integrated into a de-escalation trial.

TERTIARY OBJECTIVES:

I. To evaluate pathologic/histologic appearance of tumor after induction chemotherapy and after CRT.

II. Translational research on blood and tissue samples. III. To profile tumors genetically and immunologically in order to assess in a descriptive manner genetic or immunological features characteristic of clinical behavior.

OUTLINE:

INDUCTION CHEMOTHERAPY: All patients receive paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) over 60 minutes on days 1, 8, and 15 and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are then assigned to 1 of 3 treatment groups based on response to induction chemotherapy.

GROUP A (LOW-DOSE ARM): Patients undergo radiation therapy once daily for 5 weeks.

GROUP B (INTERMEDIATE-DOSE ARM): Patients receive hydroxyurea orally (PO) twice daily (BID) on days 0-5, fluorouracil IV continuously on days 1-5, and paclitaxel IV over 60 minutes on day 1. Patients also receive low-dose radiation therapy BID on days 1-5. Treatment repeats every 14 days for 3 courses in the absence of disease progression or unacceptable toxicity.

GROUP C (STANDARD-DOSE ARM): Patients receive hydroxyurea PO BID on days 0-5, fluorouracil IV continuously on days 1-5, and paclitaxel IV over 60 minutes on day 1. Patients also receive standard-dose radiation therapy BID on days 1-5. Treatment repeats every 14 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.*

*NOTE: At the discretion of the principal investigator (PI), patients may receive cisplatin IV over 1-3 hours every 3 weeks during radiation therapy instead of paclitaxel and undergo daily radiation therapy.

After completion of study treatment, patients are followed up for 30 days, every 3 months for 1 year, every 6 months for 2 years, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed HPV-positive squamous cell carcinoma
* HPV testing must follow the following criteria

  * HPV testing using an E6/E7 based assay is preferred, and does not require any validation (e.g. HPV in situ hybridization [ISH] or HPV E6/E7 polymerase chain reaction [PCR])
  * For oropharyngeal tumors p16 immunohistochemistry (IHC) positivity is sufficient to enroll and initiate treatment (p16 IHC interpretation to follow guidelines by Jordan/Lingen et al 2012); it is recommended that p16 IHC positivity is validated at a later point (during or after treatment) using an E6/E7 based test at the University of Chicago and provided slides will be used
  * For non-operative (OP) tumors accurate HPV testing (i.e. ISH, or E6/E7 based testing) is required for enrollment and treatment initiation
* Availability of >= 10 unstained 5 micron slides
* Patients with American Joint Committee on Cancer (AJCC) (7th edition, 2010) nodal stage N2 or N3 or a T4 primary tumor
* The primary and nodal involvement must be assessable on clinical exam (mucosal and lymph node exam)
* The primary and nodal involvement must have been defined bi- or uni-dimensional measurements measurable by RECIST
* No previous radiation or chemotherapy for a head and neck cancer
* No surgical resection for a head and neck cancer within 8 weeks of enrollment (although lymph node biopsy including excision of an individual node with presence of residual nodal disease, or surgical biopsy of the tumor is acceptable)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky >= 70%)
* Leukocytes >= 3000/mm^3
* Platelets >= 100,000/mm^3
* Absolute neutrophil count >= 1,500
* Hemoglobin > 9.0 gm/dL
* Albumin > 2.9 gm/dL
* Total bilirubin =< 1.5 mg/dl
* Creatinine clearance > 45 mL/min (or serum creatinine [SCr] =< 1.5 mg/dL), normal within 2 weeks prior to start of treatment
* The standard Cockcroft and Gault formula or the measured glomerular filtration rate must be used to calculate creatinine clearance (CrCl) for enrollment or dosing
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 X upper limit of normal (ULN)
* Alkaline phosphatase =< 2.5 X ULN
* Patients must sign a study-specific informed consent form prior to study entry; patients should have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Unequivocal demonstration of distant metastases (M1 disease)
* Intercurrent medical illnesses which would impair patient tolerance to therapy or limit survival; including but not limited to ongoing or active infection, immunodeficiency, symptomatic congestive heart failure, pulmonary dysfunction, cardiomyopathy, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance
* Pregnant and nursing women are excluded; men and women of child-bearing potential are eligible but must consent to using effective contraception during therapy and for at least 3 months after completing therapy; women with child-bearing potential must have a negative serum or urine beta-human chorionic gonadotropin (B-hCG) pregnancy test at screening
* Other coexisting malignancies or malignancies diagnosed within the previous 3 years no evidence of disease for at least 3 years; exceptions to this include non-melanoma skin cancer, cervical cancer in situ, well differentiated thyroid cancer or prostate cancer; other cancers that per assessment of the PI are not prognosis limiting can be allowed after review by the PI
* Prior surgical therapy other than incisional or excisional biopsy and organ-sparing procedures such as debulking of airway-compromising tumors or neck dissection in a patient with an unknown primary tumor; residual tumor is required for enrollment on study
* Patients receiving other investigational agents
* Peripheral neuropathy >= grade 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-09-22 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Seiwert TY, Foster CC, Blair EA, Karrison TG, Agrawal N, Melotek JM, Portugal L, Brisson RJ, Dekker A, Kochanny S, Gooi Z, Lingen MW, Villaflor VM, Ginat DT, Haraf DJ, Vokes EE. OPTIMA: a phase II dose and volume de-escalation trial for human papillomavirus-positive oropharyngeal cancer. Ann Oncol. 2019 Feb 1;30(2):297-302. doi: 10.1093/annonc/mdy522. PMID 30481287

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Radiation therapy alone, combination chemotherapy with low-dose radiation therapy, or combination chemotherapy with high-dose radiation
Period: Overall Study
Arm/Group | Single Arm
Started | 62
Completed | 61
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 62
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [54 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 56
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS), Evaluated Using RECIST Version (v) 1.1
Description: If all patients are followed for two years, the PFS rate and confidence interval will be determined based on the exact binomial distribution. Otherwise, PFS will be estimated using the Kaplan-Meier method and a (large-sample) one-sided 90% confidence interval will be derived for the PFS rate at two years to test the non-inferiority hypothesis. Median PFS will be estimated as described in Brookmeyer and Crowley.
Time Frame: Time from enrollment until disease progression or death from any cause, assessed at 2 years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 62
percentage of participants | 94.5 [88 to 96]

2. Secondary Outcome: Rate of Pathologic Complete Response (PCR) on Post Treatment Biopsy/Surgery, Evaluated Using RECIST v1.1
Description: Pathologic response rates will be determined and 95% confidence intervals obtained using the exact binomial distribution.
Time Frame: Up to 8 weeks after completion of CRT
Population: Ten missing values
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 52
percentage of participants | 90 [79 to 97]

3. Secondary Outcome: Clinical Complete Response by Computerized Tomography (CT) & Magnetic Resonance Imaging (MRI) Only
Description: Clinical response rates will be determined and 95% confidence intervals obtained using the exact binomial distribution.
Time Frame: Up to 5 years
Population: one missing value
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 61
percentage of participants
  complete response | 13 [5.8 to 24]
  Partial Response | 80 [68 to 89]
  Stable Disease | 13 [5.8 to 24]

4. Secondary Outcome: Overall Survival
Description: Overall survival rate
Time Frame: From the date of registration to the date of death or date of last patient contact if censored, assessed up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 62
percentage of participants | 87 [66 to 95]

5. Secondary Outcome: Cancer-specific Survival
Description: Overall Cancer-specific survival rate. Patients dying from non-cancer related causes will be censored at the time of death.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 62
percentage of participants | 95 [85 to 98]

6. Secondary Outcome: Rates of Acute Toxicity, Determined by Incidence of Mucositis, Xerostomia, Anorexia, Weight Loss, Dermatitis and G-tube Placement
Description: Toxicity rates will be summarized by type of toxicity, grade, and attribution. The incidence of acute (mucositis, xerostomia, anorexia, weight loss, dermatitis and G-tube placement) toxicities will be estimated along with 95% confidence intervals. Toxicity criteria of the Common Toxicity Criteria (CTC) and the Radiation Therapy Oncology Group (RTOG) will be used to determine grades. General CTC grade definitions: 0 = No adverse event or within normal limits; 1 = Mild adverse event; 2 = Moderate adverse event; 3 = Severe and undesirable adverse event; 4 = Life-threatening or disabling adverse event; 5 = Death related to adverse event. For Mucous, 3 = Confluent fibrinous, mucositis / may include severe pain requiring narcotic; 4 = Ulceration, hemorrhage or necrosis. For neutropenia, 3 = Neutrophils 0.5 - < 1.0; 4 = Neutrophils < 0.5 or sepsis.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 62
participants
  Grade 3+ mucositis | 35
  Grade 3+ dermatitis | 12
  grade 3+ neutropenia | 29
  grade 3+ Anorexia | 5

7. Secondary Outcome: Rates of Late Toxicity, Determined by Incidence of Xerostomia, Dental Decay, Osteroradionecrosis, G-tube Dependency, Tracheostomy Placement and Dysphagia
Description: Toxicity rates will be summarized by type of toxicity, grade, and attribution. The incidence of late-term (xerostomia, dental decay, osteroradionecrosis, G-tube dependency, speech abnormalities, tracheostomy placement and dysphagia) toxicities will be estimated along with 95% confidence intervals.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 62
participants
  G-tube dependence | 18
  Dysphagia | 18

8. Other Pre Specified Outcome: Histologic Appearance of Post-induction Tumor Tissue
Description: Results of pathology/histologic review of post induction biopsy specimens will be descriptive and summarize in tabular format.
Time Frame: Up to 3 months post-treatment
Population: zero analyzed because no data was collected
Arm/Group | Single Arm
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Histologic Appearance of Post-CRT Tumor Tissue
Description: as for outcome 8
Time Frame: Up to 3 months post-treatment
Population: zero analyzed because no data was collected
Arm/Group | Single Arm
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Changes in Reactive T Cells
Description: Changes in reactive T cells over time will be assessed using mixed effects models and simple paired t-tests.
Time Frame: Baseline to up to 2 months after radiation therapy
Population: zero analyzed because no data was collected
Arm/Group | Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 5 years
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 5/62
Serious Adverse Events (participants affected / at risk) | 5/62
Other Adverse Events (participants affected / at risk) | 60/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=62)
Abdominal pain (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 2
Neutrophil count decreased (Investigations) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=62)
Acute kidney injury (Renal and urinary disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 11
Alanine aminotransferase increased (Investigations) | 13
Alopecia (Skin and subcutaneous tissue disorders) | 6
Anemia (Blood and lymphatic system disorders) | 24
Anorexia (Metabolism and nutrition disorders) | 48
Anxiety (Psychiatric disorders) | 12
Aspartate aminotransferase increased (Investigations) | 9
Atrial fibrillation (Cardiac disorders) | 4
Blurred vision (Eye disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Constipation (Gastrointestinal disorders) | 51
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Dermatitis radiation (Injury, poisoning and procedural complications) | 45
Diarrhea (Gastrointestinal disorders) | 30
Dizziness (Nervous system disorders) | 5
Dry mouth (Gastrointestinal disorders) | 44
Dysgeusia (Nervous system disorders) | 52
Dysphagia (Gastrointestinal disorders) | 18
Ear pain (Ear and labyrinth disorders) | 4
Edema limbs (General disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15
Esophageal pain (Gastrointestinal disorders) | 10
Eye disorders - Other, specify (Eye disorders) | 4
Fatigue (General disorders) | 60
Fever (General disorders) | 19
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6
Headache (Nervous system disorders) | 9
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 4
Injury, poisoning and procedural complication (Injury, poisoning and procedural complications) | 4
Insomnia (Psychiatric disorders) | 10
Lymphedema (Vascular disorders) | 9
Mucosal infection (Infections and infestations) | 6
Mucositis oral (Gastrointestinal disorders) | 56
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9
Nausea (Gastrointestinal disorders) | 56
Neck edema (General disorders) | 4
Neutrophil count decreased (Investigations) | 36
Oral pain (Gastrointestinal disorders) | 21
Pain (General disorders) | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 15
Peripheral sensory neuropathy (Nervous system disorders) | 31
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 13
Platelet count decreased (Investigations) | 36
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 17
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 5
Skin ulceration (Skin and subcutaneous tissue disorders) | 7
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6
Thromboembolic event (Vascular disorders) | 6
Vomiting (Gastrointestinal disorders) | 24
Weight loss (Investigations) | 25
White blood cell decreased (Investigations) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT02258659/Prot_SAP_000.pdf